CLINICAL TRIAL: NCT04547842
Title: Mirtazapine Versus Dexamethasone in Preventing Postoperative Nausea and Vomiting After Lap Cholecystectomy a Comparative Study
Brief Title: Mirtazapine Versus Dexamethasone in Preventing Postoperative Nausea and Vomiting
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Rania Maher Hussien, MD, Lecturer of Anaesthesia and intensive care, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: FMASU R 48 / 2020
Record Dates: First submitted 2020-09-08; First posted 2020-09-14 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Post Operative Nausea and Vomiting
MeSH Terms: conditions — Vomiting | interventions — Mirtazapine; Dexamethasone

STUDY DESIGN:
Intervention Model Description: patients will be randomly divided into 2 equal groups; The M(Mirtazapine) group:(n=45) each patient will receive an oral disintegrating tablet (ODT) of mirtazapine 30 mg with sips of water and 100 ml 0.9% sodium chloride (IVI) over 15 min as a placebo 1 h preoperatively.
  The D (Dexamethasone) group: (n=45) each patient will receive a placebo tablet identical to Mirta tablet orally with sips of water and Dex 8 mg ampoule diluted in 100 ml 0.9% NS IVI over 15 min, 1 h preoperatively
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Randomization will be done using computer-generated number table of random numbers in a 1:1 ratio in opaque and sealed envelope (SNOSE). The assigned treatment will be written on a card and sealed in opaque envelopes consecutively numbered. These envelopes will be opened just immediately before administering the medication in the patient's room.
  The study drugs will be prepared by the hospital pharmacy and the patients, follow-up will be conducted by an anaesthesia resident who is not involved in any other part of the study.The patients and the investigators who collected the data will be blinded to the patient's group
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group M: patients receive Mirtazapine (Active Comparator): the patient will receive an oral disintegrating tablet (ODT) of mirtazapine 30 mg with sips of water and 100 ml 0.9% sodium chloride (normal saline [NS]) (IVI) over 15 min as a placebo 1 h preoperatively
  Interventions: Drug: Mirtazapine 30 MG
- Group D: patients receive Dexamethasone (Active Comparator): the patient will receive a placebo tablet identical to Mirta tablet orally with sips of water and Dex 8 mg ampoule diluted in 100 ml 0.9% NS IVI over 15 min, 1 h preoperatively.
  Interventions: Drug: Dexamethasone

INTERVENTIONS:
Drug: Mirtazapine 30 MG — mirtazapine is given in arm M to prevent PONV
  Other Names: Remeron
  Arms: Group M: patients receive Mirtazapine
Drug: Dexamethasone — Dexamethasone is given in arm D to prevent PONV
  Other Names: Decadrone
  Arms: Group D: patients receive Dexamethasone

SUMMARY:
Mirtazapine is a noradrenergic and specific serotonergic antidepressant. Its antagonist at the 5HT3 receptor may help to prevent nausea and vomiting. The use of mirtazapine in the management of nausea and vomiting has been reported in the literature, both for treatment and premedication.

Dexamethasone, possesses analgesic, anti-inflammatory, immune-modulating, and antiemetic effects. Dexamethasone was reported to be effective in preventing nausea and vomiting in patients receiving cancer chemotherapy. It has also been shown to be effective in reducing nausea and vomiting after open and laparoscopic surgical procedures.

In this randomized controlled trial, we will compare the effectiveness of both drugs in preventing PONV in laparoscopic cholecystectomy surgery.

DETAILED DESCRIPTION:
this double-blinded randomized study will be conducted at Ain-Shams university hospitals. Patients are aged 21-60 years and body weight 60-100 Kg of the American Society of Anaesthesiologists (ASA) physical status I or II scheduled for laparoscopic cholecystectomy under general anesthesia will be enrolled in this study., patients will be randomly divided into 2 equal groups; The M(Mirtazapine) group:(n=45) each patient will receive an oral disintegrating tablet (ODT) of mirtazapine 30 mg with sips of water and 100 ml 0.9% sodium chloride (normal saline [NS]) (IVI) over 15 min as a placebo 1 h preoperatively.

The D (Dexamethasone) group: (n=45) each patient will receive a placebo tablet identical to Mirta tablet orally with sips of water and Dex 8 mg ampoule diluted in 100 ml 0.9% NS IVI over 15 min, 1 h preoperatively.

standard monitoring in the form of (ECG, pulse oximeter, NIBP, peripheral temperature monitoring) will be attached to all patients and capnography will be connected after intubation. baseline measures will be recorded, and subsequent values will be recorded every 15 min. Patients will be observed for 24 hours postoperative. And the following will be recorded; Time to awakening (time from the end of anesthesia until the patients opened their eyes on command) and Time to the first analgesia. Patients´ vital data (BP, HR, RR, O2 saturation) will be monitored every 15 minutes for the first postoperative hour, then every 4 hours. Postoperative pain will be assessed every 4 hours with a 10-cm visual analog scale VAS (0=no pain to 10=most severe pain) score. The incidence of occurrence of postoperative Nausea and vomiting will be evaluated every 4 hours on a two-point verbal scale (0, none; 1, nausea or vomiting). The severity of nausea and vomiting will be assessed using a verbal numerical rating scale from 0 = no nausea/ vomiting and 10 = nausea/ vomiting as bad as it could be.The complete response is defined as no nausea, no vomiting, and no antiemetic medication during a 24-h postoperative period

ELIGIBILITY:
Inclusion Criteria:

* ASA physical status I or II
* body weight 60-100 Kg
* scheduled for laparoscopic cholecystectomy under general anaesthesia

Exclusion Criteria:

* Patient's refusal to participate in the study,
* Obesity with body mass index (BMI) >35 kg/m2,
* Physical status: ASA III or above,
* Patients with a history of PONV, motion sickness, or major systemic diseases
* Patients who received an antiemetic drug within 48 h before surgery,
* Patients facing liver or kidney problems with a high level of BUN or serum creatinine,
* A history of allergy to the study drugs.
* Pregnant, lactating, or menstruating patients

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2023-07-28 (Actual); Study Completion 2023-07-30 (Actual)

PRIMARY OUTCOMES:
the incidence and severity of nausea and vomiting | 24 hours postoperative
  compare the effectiveness of Mirtazapine and Dxamethasone in decreasing the incidence of PONV

SECONDARY OUTCOMES:
occurrence of postoperative complications related to the study drugs. | 24 hours postoperative
  any drug related complication

CONTACTS AND LOCATIONS:
Overall Officials: Rania Hussien, MD, Principal Investigator — Lecturer of Anaesthesia, Ain Shams University
Locations (1):
- Ain Shams University, Cairo, Abassia, Egypt